CLINICAL TRIAL: NCT00456404
Title: Effect of Peppermint Water on Prevention of Nipple Crack in Lactating Primiparous Women: a Randomized Controlled Trial
Brief Title: Effect of Peppermint Water on Breast Crack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tabriz University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 85-2
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2004-03

CONDITIONS: Breast Diseases
Keywords: peppermint water; nipple crack; lactating women
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: peppermint water

SUMMARY:
To evaluate the effectiveness of a topical preparation of peppermint water in comparison with that of expressed breast milk for the prevention of nipple cracks in primiparous breastfeeding women.

DETAILED DESCRIPTION:
One hundred and ninety-six primipara participants, who are breastfeeding after delivery at 38 or more week gestation, were assigned randomly to 2 groups, with one of 2 regimens (peppermint water, an old household remedy, and no treatment only using breast milk) to right and left sides. Each group was followed for a maximum of 3 visits within 14 days and until the 6 weeks postpartum by telephone call. The aerial parts of Mentha piperita were purchased from Hakim Momen Tabrizi Company, and the identity was confirmed by morphological characterization in comparison with the herbarium specimen retained in the School of Pharmacy, Tabriz University of Medical Sciences. Also, a voucher specimen has been generated in that herbarium.

ELIGIBILITY:
Inclusion Criteria:

* New mothers with healthy term infants (38 weeks gestation or more) are eligible for recruitment into the study. The sample of breastfeeding mothers were collected in two cohorts according delivery type. Each group consisted of 98 primipara mothers.

Exclusion Criteria:

* Mothers who didn't plan to use peppermint water
* Discharged before an interview or had preterm delivery
* Postpartum fever
* Breast infection
* Nipple abnormalities
* Age less than 18 years
* Twins
* Taking medications at night
* Mothers who didn't have telephone line, and who were illiterate.
* Infants who used bottle-feeding or pacifier, or who had mouth infection, or an abnormal short frenulum.

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 196
Dates: Start 2005-02; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome that the study was designed to evaluate: the presence and severity of sore nipples, nipple pain.
The time at which the outcome is measured: nipple and areola cracks, and pain at days 4, 8, 14.

SECONDARY OUTCOMES:
The frequency and duration of breastfeeding at days 4, 8, 14 and the number of mothers who continued feeding at week 6 was used as the secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Manizheh Sayyah Melli, MD, Study Director — Tabriz University of Medical Sciences